CLINICAL TRIAL: NCT02114086
Title: Prospective Observational Study for Intraoperative Radiotherapy (IORT) of the Breast as a Boost
Brief Title: IORT-Boost-Study, Prospective Observational Study for Intraoperative Radiotherapy of the Breast as a Boost
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kantonsspital Münsterlingen (Other)
Responsible Party: Sponsor
Other Study IDs: ROKSM 01/12; KMünsterlingen (Other: KMünsterlingen)
Record Dates: First submitted 2013-09-04; First posted 2014-04-15 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Adverse Effect of Radiation Therapy
Keywords: Observational Study; intraoperative Radiation of Breast Cancer; early and late effects of radiation; cosmesis and quality of life
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer: observation of intraoperative radiotherapy

SUMMARY:
In this study the investigators observe the investigation, whether the new method for Boost-Irradiation with the Intrabeam Device of Zeiss Germany influences local recurrence, acute and late effects of Radiotherapy, overall survival, quality of life and cosmesis.

ELIGIBILITY:
Inclusion Criteria:

* women with histologically proven unifocal ductal-invasive or other histology of breast-cancer, size of tumor < or = 3.5 cm
* written informed consent
* ability to cooperate
* full legal capability

Exclusion Criteria:

* missing written informed consent
* lack of compliance

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women with breast cancer breast-conserving therapy
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
number of Participants with local recurrence histologically proven | up to 10 years
  Recurrence of breast cancer proven by histology

SECONDARY OUTCOMES:
observation of acute and late effects of Radiotherapy | up to 10 years
  acute effects of Radiotherapy are assessed by Common Toxicity Criteria for Adverse Effects (CTCAE Version 4.0) and late effects of Radiotherapy are assessed by Late Effects Normal Tissue Subjective Objective Management Analysis (LENT-SOMA)
Overall survival | up to 10 years
  The number of Patients who died is assessed.
Quality of life | up to 10 years
  Quality of life is assessed by European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaires (QLQ) cancer modul (C30) EORTC-QLQ-C30 version 3.0 and breast cancer modul (BR23) EORTC-QLQ-BR23
Cosmesis | up to 10 years
  Cosmesis is assessed by Photographs and evaluated automatically.

OTHER OUTCOMES:
observation of influence of smoking | up to 10 years
  Patients are asked how many cigarettes they smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Reuter, Dr. med., Study Director — Kantonsspital Münsterlingen
Locations (1):
- KMünsterlingen, Münsterlingen, Thurgau, Switzerland

REFERENCES:
- [Background] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015